CLINICAL TRIAL: NCT03495115
Title: Comparing Restriction Spectrum Imaging (RSI) to Conventional and Abbreviated Breast MRI for Breast Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Radiological Society of North America (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Vandana Dialani, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 17-552
Record Dates: First submitted 2018-04-04; First posted 2018-04-11 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- SCREENING MRI (Active Comparator): Standard MRI procedure will be used.
  Interventions: Device: MRI
- SCREENING MG BI-RADS 4/5 (Experimental): * RSI is a DWI sequence with a built in distortion-correction technique that can be applied to any diffusion technique using echo planar imaging acquisition.
  * RSI will be performed using pulsed-field gradient, spin-echo, echo planar imaging with "multi-shell" diffusion data .
  * The b0 images will be collected in both the forward and reverse phase encoding directions to allow for post-processing correction of spatial distortion from magnetic field.
  Interventions: Device: RSI

INTERVENTIONS:
Device: MRI — A MRI uses a strong magnet to produce detailed pictures of the inside of your body.
  Arms: SCREENING MRI
Device: RSI — RSI is a technique that aims to improve the pictures produced during a MRI exam.
  Arms: SCREENING MG BI-RADS 4/5

SUMMARY:
This study is looking at a breast cancer screening technique, restriction spectrum imaging (RSI), as a possible alternative to the breast Magnetic Resonance Imaging (MRI) used by most healthcare professionals.

The technique involved in this study is:

-Restriction Spectrum Imaging (RSI)

DETAILED DESCRIPTION:
The primary purpose of this research study is to measure RSI's ability to diagnose breast cancer in comparison to standard breast MRIs.

RSI is a technique that has been shown to address the limitations of certain types of MRI exams used to make images of the prostate and brain. RSI is not a FDA-approved technique for screening, but is a type of advanced diffusion technique and diffusion weighted imaging is used as a part of the standard breast MRI. RSI has been shown to improve tumor detection in prostate and brain. For example, a recent pilot study in prostate showed that adding RSI improved the ability to find a certain stage of prostate cancer in comparison to an MRI without the use of the RSI technique. By comparing RSI's ability to diagnose breast cancer, future clinical testing can determine whether RSI is a more efficient way to screen for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 will consist of women who present for screening breast MRI:

  * Age >= 18
  * Female
  * Asymptomatic for breast disease
  * Presenting for routine breast cancer screening with MRI
* Group 2 will consist of women who presented for a screening mammogram (2D or 3D tomosynthesis) AND who have had a biopsy recommended after diagnostic workup:

  * Age >= 18
  * Female
  * Asymptomatic for breast disease
  * Presenting for routine breast cancer screening with mammogram (2D or 3D tomosynthesis) and/or ultrasound
  * Biopsy recommended after subsequent diagnostic workup (BI-RADS 4 or 5)

Radiologist Reader Participant

Inclusion Criteria

* Must have clinical experience in interpreting breast MRI.
* Must have interpreted at least 10 breast MRI exams with RSI interpretation.

Exclusion Criteria:

-Known or suspected renal insufficiency, rendering the participant unable to safely receive intravenous contrast based on institutional clinical protocol.

Renal insufficiency for the purposes of exclusion includes any of the following:

* Failed Chokye questionnaire
* Known history of end stage renal disease with EGFR<30 mL/min/1.73m2
* Point of care (POC) measure of creatinine clearance (eGFR) prior to obtaining the MRI <35. We will perform this POC test as needed per institutional policy for routine MRI if: (a) no creatinine result is available in the OMR within 30 days of the MRI exam, (b) the patient is > 60 years old, or (c) the patient is on hydroxyurea.

  * History of adverse or allergic-like reaction to gadolinium MRI intravenous contrast, rendering the participant unable to safely receive intravenous contrast based on institutional clinical protocol.
  * Presence of MRI unsafe devices or objects which would make having an MRI unsafe, as per institutional clinical protocol. MRI unsafe devices or objects for the purposes of exclusion include but are not limited to certain intracranial aneurysm clips, cardiac pacemaker, and implantable defibrillator devices, metallic heart valve, or coronary artery stents, breast tissue expanders, bio or neurostimulators, pellets and bullets, ocular implants and devices, otologic and cochlear implants. Other devices or metallic objects may be deemed unsafe for MRI at the radiologist's discretion.
  * Unable to tolerate exam (i.e., secondary to untreatable claustrophobia, positioning constraints/unable to lie prone).
  * Body weight exceeds that allowable by the MRI table.
  * Breast biopsy or surgical intervention planned before the test RSI-MRI in this study.
  * Breast implants (silicone or saline).

    8. Nursing or thinks she may be or is pregnant, as gadolinium contrast-enhanced MRI is unsafe. We will perform a pregnancy test as needed per institutional policy for routine breast MRI. Per institutional clinical protocol, all females of childbearing potential who are uncertain if they are pregnant or think they are pregnant must have a blood test or urine study within 2 weeks prior to the MRI exam to rule out pregnancy. A female of childbearing potential is any woman, regardless of sexual orientation or prior tubal ligation, who:
  * Has not had a hysterectomy or bilateral oophorectomy OR
  * Has not been naturally post-menopausal for at least 2 years (i.e., has had menses at any time in the preceding 2 years

Radiologist Reader Participant

-None.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of breast restriction spectrum imaging (RSI) in comparison to conventional breast MRI | 2 years
  We will test the non-inferiority of RSI compared to DCE-MRI using ROC curves created for the BI-RADS score, based on the reader study.

SECONDARY OUTCOMES:
Diagnostic accuracy of RSI compared to that of abbreviated MRI (Ab-MRI) in breast cancer screening | 2 years
  We will test the non-inferiority of RSI compared to Ab-MRI using ROC curves created for the BI-RADS score, based on the reader study.

CONTACTS AND LOCATIONS:
Overall Officials: Vandana Dialani, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No